CLINICAL TRIAL: NCT02307487
Title: Evaluation of the Safety of Pre-TURBT Intravesical Instillation of Escalating Doses of TC-3 Gel Mixed With Mitomycin C (MMC) in Non-muscle Invasive Bladder Cancer (NMIBC) Patients
Brief Title: Safety of Pre-TURBT Intravesical Instillation of Escalating Doses of TC-3 Gel and MMC in NMIBC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-BC-10
Record Dates: First submitted 2014-10-28; First posted 2014-12-04 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Bladder Cancer; Neoplasms; Urinary Bladder Diseases; Urologic Diseases
Keywords: TC-3 Gel; MMC; NMIBC; Non Muscle Invasive Bladder Cancer; Hydrogel Reverse thermal gelation; Drug retention; Urinary Bladder Neoplasms; Urologic Neoplasms; Urinary Bladder Diseases; Urologic Diseases
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms; Urinary Bladder Diseases; Urologic Diseases; Non-Muscle Invasive Bladder Neoplasms; Urologic Neoplasms | interventions — Gels; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort A2 (Experimental): 120 mg MMC in 90ml gel
  Interventions: Drug: 120 mg MMC in 90ml gel
- Cohort B2 (Experimental): 140 mg MMC in 90ml gel
  Interventions: Drug: 140 mg MMC in 90ml gel
- Cohort C2 (Experimental): 160 mg MMC in 90ml gel
  Interventions: Drug: 160 mg MMC in 90ml gel
- Cohort A (Experimental): 120 mg MMC in 60ml gel
  Interventions: Drug: 120 mg MMC in 60ml gel
- Cohort B (Experimental): 140 mg MMC in 60ml gel
  Interventions: Drug: 140 mg MMC in 60ml gel
- Cohort C (Experimental): 160 mg MMC in 60ml gel
  Interventions: Drug: 160 mg MMC in 60ml gel

INTERVENTIONS:
Drug: 120 mg MMC in 90ml gel — 120 mg of Mitomycin C mixed with 90 ml UroGen's TC-3 gel
  Other Names: Mitomycin C
  Arms: Cohort A2
Drug: 140 mg MMC in 90ml gel — 140 mg of Mitomycin C mixed with 90 ml UroGen's TC-3 gel
  Other Names: Mitomycin C
  Arms: Cohort B2
Drug: 160 mg MMC in 90ml gel — 160 mg of Mitomycin C mixed with 90 ml UroGen's TC-3 gel
  Other Names: Mitomycin C
  Arms: Cohort C2
Drug: 120 mg MMC in 60ml gel — 120 mg of Mitomycin C mixed with 60 ml UroGen's TC-3 gel
  Other Names: Mitomycin C
  Arms: Cohort A
Drug: 140 mg MMC in 60ml gel — 140 mg of Mitomycin C mixed with 60 ml UroGen's TC-3 gel
  Other Names: Mitomycin C
  Arms: Cohort B
Drug: 160 mg MMC in 60ml gel — 160 mg of Mitomycin C mixed with 60 ml UroGen's TC-3 gel
  Other Names: Mitomycin C
  Arms: Cohort C

SUMMARY:
A prospective, open label, modified 3+3 dose escalation study. This dose-escalation study is designed to carefully assess the safety of successive cohorts of patients (3 patients/cohort), each cohort treated with a fixed dose of TC-3 and MMC Intravesical instillations.

DETAILED DESCRIPTION:
A prospective, open label, modified 3+3 dose escalation study. This dose-escalation study is designed to carefully assess the safety of successive cohorts of patients. A total of 10 patients will be treated in the first cohort with 120mg MMC-TC-3 Gel unless DLT is reached in more than 1/3 of the patients in the cohort. The next cohorts will have 3 patients/cohort, each cohort treated with a fixed dose of TC-3 and MMC Intravesical instillations. Since data is already available for 40 and 80 mg MMC in TC-3 gel, the initial cohort is 120mg MMC mixed with of 60 mL TC-3. Subsequent cohorts will be given dose levels of 140mg & 160mg MMC mixed with 60 mL TC-3. Thus, if 160mg MMC mixed in 60ml TC-3 will be found to be safe and tolerable, no higher doses will be further explored at this stage.

If 120 mg MMC in 60 ml TC-gel (2 mg/ml) is found to be intolerable, higher concentrations will not be tested. Instead, a dose of 120 mg in 90 cc TC gel and a subsequent doses of 140 and 160 mg MMC in 90 cc TC gel will be tested in the same dose escalating manner. This will allow testing similar doses at lower concentrations (up to 1.78 mg/ml) but with a longer dwell time due to the larger volume of TC-gel.

Dose escalation is to be halted when the maximum tolerated dose (MTD) will be reached; MTD is defined as one dose level below which dose limited toxicity (DLT) is Any adverse event (AE) related to TC-3+MMC and qualified per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) as grade 3 or 4 will be evaluated by board of 2 independent physicians to determine if it qualifies as DLT based on the known safety profile of MMC. If the NCI grade will not apply, the adverse event to be graded as mild, moderate, or severe.

If one of the three patients in a cohort experienced a DLT, three more patients will be added to the cohort for AE confirmation, only if 3 patients from the given cohort will experienced DLT, the MTD will be reached If no further DLTs are observed in the cohort, the three patients will be enrolled in the next successive cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older.
* Patient has signed Informed Consent Form and is willing and able to abide by the protocol.
* Patients diagnosed with Low Grade (LG) or High grade (HG) NMIBC.
* No active urinary tract infection as confirmed by urine culture.
* If the patient is a female of childbearing potential, she is using two acceptable & effective methods of contraception, until 6 months post treatment
* A negative serum pregnancy test at screening for female patient with childbearing potential
* If the patient is a male he should use a condom during intercourse, for at least 48 hours post each instillation.
* If the patient is a male that has a partner that is a female of childbearing potential, he should be advised to use two acceptable & effective methods of contraception until 6 months post treatment.

Exclusion Criteria:

* Tumor located in prostatic urethra (for male patient) or in the bladder diverticulum.
* Prior or required pelvic radiotherapy.
* Systemic chemotherapy within 1 year prior the screening.
* Pregnant or breastfeeding female patient.
* Treatment of bladder cancer with BCG within the last 12 months prior to screening visit . Exception: For patient that had BCG treatment within 6-12 months prior to screening visit and are not symptomatic, the patient may enroll at the investigator discretion.
* Treatment (full course) with intravesical chemotherapy within the 3 months, prior to screening visit.
* Contraindication to MMC treatment as per investigator determination, or known sensitivity to MMC or TC-3 ingredients.
* The patient has a known current urinary retention which requires intermittent catheterization to empty the bladder.
* The patient has a bleeding disorder or a screening platelet count <100X109/L.
* The patient has screening hemoglobin <10g/dL OR white blood cells < 4000 mm3.
* GFR<30
* Hepatic values exceeding 2 times the upper normal limit.
* The patient has a concurrent severe and/or uncontrolled medical condition (e.g., uncontrolled diabetes, compensated congestive heart failure [NYHA III and over], myocardial infarction within 6 months of screening visit, unstable or uncontrolled hypertension or an active uncontrolled infection) or psychiatric disease, which could compromise participation, compliance with scheduled visits, and/or completion of the study in the opinion of the investigator.
* The patient has a documented severe vesico-ureteral reflux or has an in-dwelling ureteral stent.
* The patient participated in an investigational interventional study within the past 90 days, prior to screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Rate of Adverse Events (AE) findings considered to be dose limiting according to the CTCAE V 4.0 | 6 weeks
Vital signs findings considered to be dose limiting according to the CTCAE V 4.0 | 6 weeks
Clinical evaluation findings considered to be dose limiting according to the CTCAE V 4.0 | 6 weeks
Lab results considered to be dose limiting according to the CTCAE V 4.0 | 6 weeks

SECONDARY OUTCOMES:
Rates of all adverse events or clinically relevant physical examination | 15 months
Vital signs and laboratory findings | 15 months
MMC maximum plasma concentration and concentration time curve during 6 hr post instillation | 15 months
Duration of MMC retention in the bladder as detected by urine MMC levels post instillation (6-7 hours) | 15 months

OTHER OUTCOMES:
Rate of patients with Complete Response (CR) to treatment | 8-10 weeks post treatment
  Complete Response (CR) rate defined as percent of patients with CR at the Primary Disease Evaluation (PDE) Visit
Rate of patients with durable Complete Response (CR) to treatment | 3, 6, 9 and 12 months post PDE visit
  Durable Complete Response (CR) rate defined as percent of patients who continue to display CR at 3, 6, 9 and 12 months following the last treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ifat Klein, PhD, Study Director — UroGen Pharma
Locations (2):
- Israel (2):
  - Wolfson Medical Center of Holon, Department of Urology, Holon
  - Meir Medical Center, Kfar Saba

REFERENCES:
- [Derived] Prasad SM, Louie MJ, Burger B, Tsurutis V, Ugwuoke N, Strauss-Ayali D. Pharmacokinetics of UGN-102, an investigational mitomycin-containing reverse thermal gel for the treatment of non-muscle invasive bladder cancer. Cancer Chemother Pharmacol. 2025 Oct 11;95(1):100. doi: 10.1007/s00280-025-04821-5. PMID 41074972
- See also: UroGen pharma official website — http://www.urogen.com/